CLINICAL TRIAL: NCT02155582
Title: A Phase I Pharmacodynamic Study of Copanlisib (BAY 80-6946) as Monotherapy in Patients With Non-Hodgkin's Lymphoma and Solid Tumors
Brief Title: Copanlisib Pharmacodynamic Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16790; 2013-004746-42 (EudraCT Number)
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Non Hodgkin Lymphoma
Keywords: Solid tumors
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — copanlisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): 0.8 mg/kg body weight and 0.4 mg/kg (not to exceed 65 mg) for the non-diabetic patients
  Interventions: Drug: Copanlisib (BAY80-6946)
- Arm 2 (Experimental): 45 mg and 60 mg for the diabetic patients
  Interventions: Drug: Copanlisib (BAY80-6946)

INTERVENTIONS:
Drug: Copanlisib (BAY80-6946) — 0.8 mg/kg body weight and 0.4 mg/kg (not to exceed 65 mg) for the non-diabetic patients;45 mg and 60 mg for the diabetic patients; Intravenous (IV) infusion over 1 hour. Dosing of copanlisib will be on Days 1, 8, and 15 of each 28 day treatment cycle.

SUMMARY:
This study aims to analyze what the study drug does to the body and its relationship to drug levels and safety after patients with advanced cancer have been treated with copanlisib in different dose groups.

ELIGIBILITY:
* Histologically confirmed diagnosis of the following NHL: follicular lymphoma all grades, lymphoplasmacytic lymphoma / Waldenström macroglobulinemia, transformed indolent lymphoma, diffuse large B-cell lymphoma, Burkitt lymphoma, mantle cell lymphoma, or peripheral T-cell lymphoma, relapsed or refractory, with 1 or more prior chemo-immunotherapy- or immunotherapy-based regimen(s) OR
* Advanced and / or refractory solid tumors with high prevalence (≥30%) of PIK3CA or PTEN alteration: Breast and uterine cancers (endometrium cancers but also non-endometrial uterine cancers), lung (squamous cell only), cervical, head and neck, prostate, and ovarian cancers
* Biopsy-accessible tumor
* Male or female patients equal 18 or more years of age
* NHL patients must have at least 1 bi-dimensionally measurable lesion according to the modified Cheson criteria. Patients with solid tumors must have at least 1 solid tumor lesion measurable by computed tomography or magnetic resonance imaging according to the Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) criteria
* Eastern Cooperative Oncology Group performance status 2 or <
* Life expectancy of at least 3 months
* Adequate bone marrow, liver, and renal functions as assessed by laboratory requirements conducted within 7 days before the first dose of study drug
* Left ventricular ejection fraction > or equal the lower limit of normal for the institution

Exclusion Criteria:

* Previous or concurrent cancer that is distinct in primary site or histology from NHL or the solid tumor, for which the patient is enrolled into this study, within 5 years before treatment start EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer, in situ breast cancer, in situ prostate carcinoma if Gleason score < or equal to 6 and prostate-specific antigen <10 ng/mL, and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor invades lamina propria)]
* Known lymphomatous involvement of the brain or leptomeningeal involvement; solid tumor patients with central nervous system (CNS) metastases if treatment completed <3 months before enrollment or lesions unstable or progressing on magnetic resonance imaging scans performed within 1 month of enrollment or unstable symptoms of the CNS metastases
* Any illness or medical condition that is unstable or could jeopardize the safety of the patient or his / her compliance in the study
* Current diagnosis of type 1 or type 2 diabetes mellitus with HbA1c < or equal to 8.5% or fasting blood glucose < or equal to 160 mg/dL

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2014-08-12 (Actual); Primary Completion 2016-10-04 (Actual); Study Completion 2017-03-16 (Actual)

PRIMARY OUTCOMES:
Maximum change from baseline in expression of pathway inhibition (pAKT) in surrogate tissue (platelet rich plasma) during copanlisib monotherapy | Baseline and approximately 2 years
Maximum change from baseline in plasma glucose during 2 cycles of copanlisib monotherapy | Baseline and after day 22

SECONDARY OUTCOMES:
AUC(0-168) of copanlisib after each copanlisib IV infusion during 2 cycles of copanlisib monotherapy | After day 22
AEs as characterized by type, frequency, severity (as graded by CTCAE) and relationship to study drug | Approximately 2 years
Maximum change from baseline in insulin during 2 cycles of copanlisib | After day 22
Maximum change from baseline in C-peptide during 2 cycles of copanlisib | After day 22
FDG PET early response (decreased SUVmax compared to baseline) after dosing with copanlisib for non-diabetic patients with detectable FDG tumor uptake at baseline | After day 22
Change from baseline in expression and / or phosphorylation of PI3K pathway proteins in paired tumor biopsies | Baseline and after day 22

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (8):
- Belgium (2):
  - Bruxelles - Brussel
  - Ghent
- France (4):
  - Caen
  - Lille
  - Nice
  - Pierre-Bénite
- United Kingdom (2):
  - Sutton, Surrey
  - London